CLINICAL TRIAL: NCT05357950
Title: A Phase IIb, Randomized, Multi-Center, Multinational, Prospective, Double-Blind, Placebo-Controlled Study, With an Open Label Extension, to Evaluate Safety, Tolerability and Efficacy of PrimeC in Subjects With ALS
Brief Title: A Phase IIb, Multi-Center, Multinational, Double-Blind, Placebo-Controlled Study, With an Open Label Extension, to Evaluate Safety, Tolerability and Efficacy of PrimeC in Subjects With ALS
Acronym: PARADIGM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroSense Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NST003
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrimeC (Active Comparator): 2 tablets of PrimeC administered twice daily (4 tablets a day), at a daily dose of 1496 mg
  Interventions: Drug: PrimeC
- Placebo (Placebo Comparator): 2 tablets of Placebo administered twice daily (4 tablets a day). Placebo tablets are matched in size, color and taste.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PrimeC — Ciprofloxacin and celecoxib combination extended release formulation
  Arms: PrimeC
Drug: Placebo — Placebo matches active drug in size, color and taste
  Arms: Placebo

SUMMARY:
69 subjects with ALS will be enrolled in the study and randomized at a 2:1 ratio to receive the study drug or placebo tablets. Randomization sequences will be in random block sizes and stratified for ENCALS risk category [high risk ≥ -4.5 vs. low risk < -4.5], and for background ALS treatment (riluzole and/or edaravone and/or sodium phenylbutyrate and/or taurursodiol) vs. no background ALS treatment.

All subjects will be administered the drug/placebo twice daily (BID), two tablets each time, for 6 months. Subjects will be allowed to receive standard of care (SOC) treatment of approved products (i.e., riluzole and edaravone). Additionally, subjects will be allowed to receive treatment with off-label sodium phenylbutyrate and taurursodiol, which are accepted for ALS treatment.

Subjects will be evaluated every 2 months for safety, tolerability (adverse events, safety laboratory, vital signs, ECG, withdrawal rates and reasons) and efficacy (e.g. biomarkers, clinical outcomes (ALSFRS-R and SVC, quality of life and survival).

All subjects who complete the 6 months dosing will be switched to the active arm for a 12-month open label extension (OLE).

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF)
2. Males or females between the ages of 18 and 75 years of age, inclusive
3. Diagnosis of familial or sporadic ALS (defined as meeting the laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the Gold Coast criteria)
4. Disease duration after first symptom (muscle weakness) less than 30 months prior to screening
5. Pre-enrollment ALSFRS-R slope from disease onset ≥ 0.3 points per month
6. ALSFRS-R at screening ≥ 25
7. Item 3 (swallowing) in ALSFRS-R ≥ 3
8. Subjects may be treated in parallel with riluzole and/or edaravone and/or sodium phenylbutyrate and/or taurursodiol; 60 days of stable use prior to enrollment is required
9. Upright slow vital capacity (SVC) ≥ 60% of predicted for age, height, weight and sex at screening according to the GLI-2012
10. 18 < BMI < 30
11. A caregiver (if one is needed)
12. Female subjects must be post-menopausal (≥ 1 year) OR sterilized, OR if of childbearing potential (i.e., females who have had their first period unless they are anatomically or physiologically incapable to become pregnant), must have a negative pregnancy test, and agree to use contraceptive drugs or devices (e.g., diaphragm plus spermicide, or oral contraceptives) for the duration of the study and 10 weeks after the last treatment dose AND require male partners to use a condom during sexual intercourse

Exclusion Criteria:

1. A past history of adverse reaction/hypersensitivity to either NSAIDs, celecoxib or fluoroquinolones, ciprofloxacin
2. Any known clinically significant abnormal gastric mucosal erosion, ulcer or tumor or/and GI disorder and/or bariatric surgery
3. Known history of clinically significant impairment of renal function (creatinine ≥ 1.5)
4. Known or suspected symptomatic congestive heart and/or coronary heart disease, previous history of myocardial infarction, uncontrolled arterial hypertension, or rhythm abnormalities requiring permanent treatment
5. Known history of QT/QTc prolongation, Torsade de pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT syndrome) and the use of concomitant medications that prolong the QT/QTc interval
6. Known or suspected diagnosis or family history of epilepsy in first degree relatives
7. Known predisposition to tendinitis
8. Known or suspected to be a poor CYP2C9 metabolizers who also uses pharmacologic agents (prescription or over-the-counter) or herbal products known or suspected to induce or inhibit CYP2C9 within 30 days before enrollment
9. Tracheostomy or percutaneous gastrostomy use
10. Presence at screening of any medically significant cardiac, pulmonary, musculoskeletal, or psychiatric illness that might interfere with the subject's ability to comply with study procedures or that might confound the interpretation of clinical safety data, including, but not limited to:

    1. Mean systolic blood pressure >160 mm Hg and/or mean diastolic blood pressure >100 mm Hg (measurements taken after a few minutes rest) that persist on 3 successive measurements taken at least 2 minutes apart
    2. NYHA Class II or greater congestive heart failure
    3. Chronic obstructive pulmonary disease or asthma requiring daily use of bronchodilator medications
    4. Poorly controlled or brittle diabetes mellitus
    5. Cognitive impairment, related to ALS or otherwise, sufficient to impair subject's ability to understand and/or comply with study procedures and provide informed consent
11. Subject who is treated with chronic aspirin or NSAIDs and is at risk if stopped. Clopidogrel is allowed and can replace Aspirin.
12. Any contraindication for ciprofloxacin and celecoxib according to the current prescribing information.
13. Female who is pregnant or breastfeeding or with intention of becoming pregnant during the course of the study.
14. Any impairment or social circumstance that, in the opinion of the Investigator, would render the subject not suitable to participate in the study.
15. Subject, or subject's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
16. Subject is participating in (or plans to participate in) any other investigational drug trial, or plans to be exposed to any other investigational agent, device and/or procedure, from 30 days prior to Screening through study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 6 months
  Treatment emergent adverse event is any medical event associated with the drug
Number of subjects who discontinued treatment prematurely | 6 months
  Number of subjects whose treatment is stopped prematurely for any reason
Number of patients who discontinued treatment prematurely due to adverse events | 6 months
  Number of patients whose treatment is stopped prematurely specifically due to adverse events
Number of patients with clinically significant abnormal laboratory values | 6 months
The mean difference between PrimeC and Placebo in serum concentration of NDE TDP-43 at month 6 | 6 months
The mean difference between PrimeC and placebo in serum concentration of NDE PgJ2 at month 6 | 6 months

SECONDARY OUTCOMES:
Change from baseline to 6 months in ALS functional rating scale - revised (ALSFRS-R) | 6 months
Change from baseline to 6 months in slow vital capacity (SVC) | 6 months
Change from baseline to 6 months in quality of life ALSSQOL-SF | 6 months
Change from baseline to 6 months in PROMIS-10 quality of life questionnaire | 6 months
Survival at 6 months of treatment | 6 months
  Overall Survival defined as time to death from any cause at 6 months of treatment
Composite survival at 6 months of treatment | 6 months
  Composite of overall survival, defined as time to death from any cause, or respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥22 h per day for ≥10 consecutive days) at 6 months of treatment
Composite survival at 6 months of treatment | 6 months
  Composite of overall survival, defined as time to death from any cause, or respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥22 h per day for ≥10 consecutive days), or time to hospitalization due to ALS-related complications at 6 months of treatment
Joint Assessment of Function and Survival after 6 months of treatment | 6 months

OTHER OUTCOMES:
Change from baseline to 6 months in the following serum biomarkers: serum ferritin, transferrin, iron, neurofilaments and exosomal LC3, Dicer, and other biomarkers evaluating the effect of PrimeC on pathophysiological mechanisms in ALS | 6 months
Effect of PrimeC versus placebo on the time to reach advanced disease stages (King's/MiToS) | 6 months
Change from baseline to 6 months in Patient-ranked order of function (PROOF) | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Lawson Health Research Institute, London, Ontario, Canada
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - IRCCS Istituti clinici Maugeri, Milan
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: Undecided